CLINICAL TRIAL: NCT04270526
Title: Minimizing Pain During Office Intradetrussor Botox Injection: A Prospective Randomized Controlled Trial Comparing Two Protocols
Brief Title: Minimizing Pain During Office Intradetrussor Botox Injection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Urogynecology Associates (Other)
Responsible Party: Principal Investigator, William D. Winkelman, Clinical Instructor, Boston Urogynecology Associates
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 037-2019
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Results first posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Overactive Bladder; Overactive Detrusor; Overactive Bladder Syndrome; Overactivity; Behavior; Urge Incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Spasm; Urinary Incontinence, Urge | interventions — AIEOP acute lymphoblastic leukemia protocol

STUDY DESIGN:
Intervention Model Description: All subjects will be randomized 1:1 at the first intervention visit to one of the two protocols using a random block design
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active treatment (Active Comparator): 50 mL 1% lidocaine + 45ml of 0.9% normal saline + 5 mL 8.4% sodium bicarbonate
  Interventions: Drug: Bicarbonate protocol
- Placebo treatment (Placebo Comparator): 50 mL 1% lidocaine + 50ml of 0.9% normal saline
  Interventions: Drug: Standard protocol

INTERVENTIONS:
Drug: Bicarbonate protocol — Intradetrussor treatment with 50 mL 1% lidocaine + 45ml of 0.9% normal saline + 5 mL 8.4% sodium bicarbonate
  Arms: Active treatment
Drug: Standard protocol — Intradetrussor treatment with 50 mL 1% lidocaine + 50ml of 0.9% normal saline
  Arms: Placebo treatment

SUMMARY:
This will be a prospective double-blinded randomized controlled trial comparing two pre-treatment protocols for patients undergoing intradetrussor botox injections to determine if a buffered lidocaine solution offers superior pain control.

DETAILED DESCRIPTION:
Lidocaine is a commonly used amide-type local anesthetic. Lidocaine exists as both a quaternary water soluble structure, and a tertiary lipid-soluble structure. Only the tertiary lipid-soluble structure can cross the lipid bilayer of a cell membrane and thereby enter a neurons axoplasm and induce the desired effect. The ionization constant of lidocaine is 7.7 which means that at a pH of 7.7, 50% of lidocaine is available in the tertiary lipid-soluble structure. At a physiologic pH between 7.35 and 7.45 only around 44% of lidocaine is in the tertiary lipid-soluble structure. However, for lidocaine to be stable in solution, it is typically formulated as a hydrochloride salt and the pH of most commercially available lidocaine solutions are at a pH of 6.09. In an acidic solution the majority of lidocaine is available in the quaternary water-soluble structure and at this pH only 2.5% of lidocaine is in the tertiary lipid-soluble structure. A Cochrane review found that increasing the pH of lidocaine prior to injection decreased pain and increased patient satisfaction perhaps because of the aforementioned pharmacokinetic principles.

Lidocaine is typically used as anesthetic for intradetrussor injections of onabotulinum toxin A for the treatment of refractory overactive bladder. In 2003, a technique for intradetrussor injections of onabotulinum toxin A was first described using only local anesthesia. At that time, the procedure involved intrauerthral lidocaine. The procedure has evolved since that time and currently many physicians utilize protocols with both utraurethral and intravesical lidocaine. At baseline intradetrusor onabotulinum toxin A injections are generally well tolerated and with reported mean VAS scores around 3.

For patients with refractory overactive bladder, the standard of care is intradetrussor onabotulinum toxin A injections. The standard protocol used by the investigators involves emptying the bladder then retrograde filling the bladder with a 1:1 mixture of 1% lidocaine normal saline. This solution remains in the bladder for approximately 15 minutes prior to injection. Given that urine is typically acidic and commercially available lidocaine solutions are similarly acidic, it is likely that only a fraction of intravesical lidocaine is in the active tertiary lipid-soluble form. The goal of this study is to determine if the investigators can improve the procedural pain of intradetrusor onabotulinum toxin A injections using a buffered solution compared to our standard solution.

After approval by the IRB, investigators will approach possible participants who are having intradetrussor botox injection for overactive bladder which is the standard of care for patients with refractory overactive bladder. If the patient meets eligibility criteria, consent forms will be signed and the patient will be randomized 1:1 to receive either our standard pretreatment regimen with 50 mL 1% lidocaine + 50ml of 0.9% normal saline or our buffered bicarbonate protocol with 50 mL 1% lidocaine + 45ml of 0.9% normal saline + 5 mL 8.4% sodium bicarbonate. The primary end point of this trial is to assess the pain scores measured on a Visual Analogue Scale (VAS) immediately following the procedure. Secondary end points include patient satisfaction, willingness to undergo repeat treatment and adverse events.

All subjects will be randomized 1:1 at the first intervention visit to one of the two protocols using a random block design . At the completion of the procedure, patients will be asked to complete a brief questionnaire about their experience. Patients will follow up in clinic for a post-void residual check two weeks after the procedure as is standard for our clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Female patient
* Primary diagnosis of overactive bladder
* Failed first and second line therapy for overactive bladder
* Planning to undergo bladder botox injections

Exclusion Criteria:

* Neurogenic bladder
* Urinary retention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Urogynecology Associates, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Treatment | Placebo Treatment
Started | 38 | 38
Completed | 36 | 37
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Treatment | Placebo Treatment | Total
Number analyzed (Participants) | 37 | 36 | 73
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 74 [67 to 78] | 71 [65 to 78] | 72 [66 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 36 | 73
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 32 | 30 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: Pain: VAS
Description: Pain on visual analog scale from 0-100 with higher scores worse
Time Frame: Immediately after the procedure
Measure: Median (Inter-Quartile Range); unit: units on a scale, 0-100
Arm/Group | Active Treatment | Placebo Treatment
Number analyzed (Participants) | 37 | 36
units on a scale, 0-100 | 25 [15 to 55] | 16 [9 to 40]

2. Secondary Outcome: Satisfaction: Likert Scale
Description: Likert scale questions assessing overall satisfaction with the procedure with responses from very 1 (dissatisfied) to 5 (very satisfied) with higher scores representing more satisfaction. We reported the percentage of participants who were satisfied we defined as a response of 4 or 5.
Time Frame: Immediately after the procedure
Measure: Number; unit: percentage of participants with 4 or 5
Arm/Group | Active Treatment | Placebo Treatment
Number analyzed (Participants) | 37 | 36
percentage of participants with 4 or 5 | 68 | 39

3. Secondary Outcome: Willingness to Undergo Repeat Procedure
Description: Likert scale questions assessing the patient's willingness to undergo a repeat procedure from very likely (1) to very unlikely (5) with five items total. We defined willingness to undergo repeat procedure as a score of 1 or 2 on the Likert scale and outcome measured was the percentage of patients who responded with a 1 or 2.
Time Frame: Immediately after the procedure
Measure: Number; unit: percentage of participants
Arm/Group | Active Treatment | Placebo Treatment
Number analyzed (Participants) | 37 | 36
percentage of participants | 72 | 65

ADVERSE EVENTS:
Time Frame: 1 hour
Arm/Group | Active Treatment | Placebo Treatment
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/37
Other Adverse Events (participants affected / at risk) | 0/37 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/26/NCT04270526/Prot_SAP_003.pdf
  • Informed Consent Form (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/26/NCT04270526/ICF_004.pdf